CLINICAL TRIAL: NCT02544399
Title: Is Golf a Sport Suited to the Female Skeleton After 60 Years? Pilot Study Evaluating the Microarchitecture 3D Carriers and Noncarriers Bones
Brief Title: Bone Microarchitecture in Women Practicing Golf
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0801092; 2008-A01265-50 (Other: AFSSAPS)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Bone Microarchitecture
Keywords: Bone microarchitecture; Playing golf; Walkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subject practicing golf and accept bone measure: Each patient will have 1 blood sample and 1 measure of bone by 3D micro-tomography
  Interventions: Other: 3D CT scan
- Subject practicing foot walk and accept bone measure: Each patient will have 1 blood sample and 1 measure of bone by 3D micro-tomography
  Interventions: Other: 3D CT scan
- Subject sedentary and accept bone measure: Each patient will have 1 blood sample and 1 measure of bone by 3D micro-tomography
  Interventions: Other: 3D CT scan

INTERVENTIONS:
Other: 3D CT scan — Measure of bone micro-architecture by 3D micro-tomography

SUMMARY:
After the age of 50, one in three women and one in eight men will experience at least one fragility fracture during the rest of their lives. It is currently recognized that physical activity has an osteogenic actions, especially when it includes the impact transmitted to the skeleton. In this context, the investigators propose a study to determine whether the regular practice of golf could be particularly beneficial for the skeleton, not only in the lower limbs, due to repeated impacts to the ground when it requires sustained walking, but also the upper limbs due to the impacts transmitted by the club at the time of striking the ball, as has been amply demonstrated with racquet sports.

DETAILED DESCRIPTION:
Each patient will have 1 blood samples and 1 measure of bone by 3D micro-tomography (3D CT Scan).These examinations and sampling will take place on 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Golfers: Regular playing golf for over 2 years at 8 to 12 hours per week recruited into golf clubs.
* Walkers: regular practice of walking for over 2 years at 8 to 12 hours per week recruited into the walking clubs.
* Sedentary: no intensive physical activity (<2 hours / week), recruited in clubs seniors.

Exclusion Criteria:

* concomitant bone disease ,
* Hip prosthesis the dominant side
* Endocrinopathy
* hypercalcemia, vitamin D deficiency, hypo- or hyper calciuria
* Active smoking (more than 5 cigarettes / day), chronic alcoholism,
* Treatments received in the previous six months and resounding on bone metabolism such growth promoters, all osteoporosis, corticosteroids.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject practicing foot walk or golf or sedentary
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bone volume / tissue volume | day 1
  Measure of Bone volume / tissue volume by the 3D CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Thierry THOMAS, MD-PhD, Principal Investigator — CHU SAINT-ETIENNE